CLINICAL TRIAL: NCT01114126
Title: Randomized, Double-blind, Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics of Neu-P11 in Subjects With Primary Insomnia
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Neu-P11 in Subjects With Primary Insomnia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Dr. Tali Nir, VP clinical and regulatory affairs, Neurim Pharmaceuticals Ltd.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Neu-P11
Record Dates: First submitted 2010-04-15; First posted 2010-04-30 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Insomnia
Keywords: Neu-P11; Insomnia; PSG; safety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — N-(2-(5-methoxy-indol-3-yl)-ethyl)-4-oxo-4H-pyran-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Neu-P11 2mg (Experimental)
  Interventions: Drug: Neu-P11
- Neu-P11 5 mg (Experimental)
  Interventions: Drug: Neu-P11
- Neu-p11 20 mg (Experimental)
  Interventions: Drug: Neu-P11
- Neu-P11 50 mg (Experimental)
  Interventions: Drug: Neu-P11
- Placebo (Placebo Comparator)
  Interventions: Drug: Neu-P11 placebo

INTERVENTIONS:
Drug: Neu-P11 — comparison of different dosages of drug
  Arms: Neu-P11 2mg; Neu-P11 5 mg; Neu-P11 50 mg; Neu-p11 20 mg
Drug: Neu-P11 placebo — comparison of different dosages
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of Neu-P11, following the administration of multiple ascending oral doses (2, 5, 20, 50 mg or matching placebo) given nightly over 2 periods of 5 days to male and female subjects with primary insomnia. In addition, the study is aimed to determine the pharmacokinetic profile of Neu-P11 after 1 and 5 days of administration and to evaluate the hypnotic effects of Neu-P11 as well as the effects on mood and memory. The study hypothesis is that Neu-P11 is safe, tolerated and have significant sleep promoting effects.

DETAILED DESCRIPTION:
The effects of four multiple ascending doses of orally administered Neu-P11 will be evaluated in a double- blind, placebo-controlled, crossover design. Following a screening visit, the recruited subjects will undergo an inclusion/habituation full night PSG screening recording in the sleep clinic to exclude subjects with sleep disorders. Eligible subjects will be divided into 2 cohorts of 12 subjects each. Following screening, each cohort will be randomised to receive Neu-P11 or placebo for a first period of 5 days and will be crossed over following at least 21 days to receive placebo or a higher dose of Neu-P11 for a second period of 5 days. Each cohort will receive a different dose of Neu-P11, chosen from 2, 5, 20 and 50 mg. The starting dose is 5 mg but a smaller dose (2 mg) is also included for the purpose of pharmacodynamic evaluation. Before proceeding from 5mg to the next higher dose safety will be evaluated based on adverse events, clinical and biological data. Subjects of Cohort A will be randomised to dose levels 2 and 3 (doses 5 and 20 mg). Subjects of Cohort B will be randomised to dose levels 1 and 4 (doses 2 and 50 mg).

ELIGIBILITY:
Inclusion Criteria:

1. Primary insomnia male or female subjects according to DSM-IV criteria (307.42) ,
2. Sleep latency of > 30 minutes and total sleep time < 6 hrs based on Sleep History Questionnaire (SHQ) and verified by the inclusion + habituation night PSG,
3. Men or women 18 to 65 years inclusive,
4. Women of childbearing potential must have a negative pregnancy test at the screening visit, on Day 1 of each treatment period, and use a reliable method of contraception during the entire study duration and for at least 3 months after study drug intake. Reliable methods of contraception are:

   * Double barrier type devices (e.g., male or female condom, diaphragm, contraceptive sponge) only in combination with a spermicide.
   * Intra-uterine devices in combination with a spermicide. Abstention, rhythm method, and contraception by the partner alone are not acceptable methods of contraception. Women not of childbearing potential are defined as postmenopausal (i.e., amenorrhea for at least 1 year), or surgically or naturally sterile.
5. Subjects must be in good health as determined by their medical history, physical examination, ECG, vital signs, standard EEG, serum biochemistry, haematology and urinalysis. A subject with clinical abnormality may be included only if the investigator or his designee considers that the abnormality will not introduce additional risk factor for the subject's health, or interfere with the study objectives,
6. Subjects who have not been using BZD and non-BZD hypnotics or melatoninergic drugs for the past 2 weeks or more prior to Screening,
7. Subjects who have not been using psychotropic treatments for the past 3 months or more prior to screening,
8. Subjects who have not been using any other non-psychotropic treatments for the past 2 weeks or more prior to Screening with the exception of occasional paracetamol intake (1 g per day),
9. Subjects having read and signed the informed consent form,
10. Subjects having a body mass index between 18 and 30 (extremes included),
11. Subjects having no documented hypersensitivity to exogenous melatonin or agonists,
12. Subjects who agree to completely refrain from alcohol, caffeine and tobacco during the institutionalisation periods,
13. Subjects able to take part in the whole study,
14. Subjects affiliated with, or beneficiary of, a social security system

Exclusion Criteria:

1. According to DSM IV, subjects belonging to the following groups are excluded: 780.59 (breathing related sleep disorder); 307.45 (circadian rhythm sleep disorder); 307.47 (dyssomnia not otherwise specified); 780.xx (sleep disorder due to general medical condition) ,
2. Subjects suffering from insomnia secondary to other causes according to SHQ,
3. Subjects with sleep disorders detected during the PSG inclusion/habituation night, such as sleep apnea/hypopnea and periodic leg movement syndrome (with arousal) (PLMI > 15 and/or AHI > 15 per hour),
4. Subjects with known chronic infections or asthma, allergies or history of severe allergy,
5. Subjects with hypertension defined as systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg according to two repeated measures in lying position within 10 min interval,
6. Subjects with hypotension defined as systolic blood pressure <90 mmHg and/or diastolic blood pressure < 45 mmHg according to two repeated measures in lying position within 10 min interval,
7. Subjects with foreseeable need of a treatment, whatever it is (including dental care), during the study period,
8. Subjects with positive drug screening for amphetamines, benzodiazepines, barbiturates, cannabis, cocaine morphine/opiates, methadone, tricyclics, methamphetamines (ecstasy) and codeine, or suspected to be drug or alcohol addicted,
9. Subjects with positive serology to human immunodeficiency virus antibodies (HIV Ab),
10. Subjects positive for Hepatitis B virus surface antigen (HBs Ag) or hepatitis C virus antibodies (HCV Ab),
11. Subjects with previous or on-going chronic or recurrent disease especially convulsive disorders or central nervous system or psychiatric disease,
12. Subjects with history of pathology likely to recur during or immediately after the study,
13. Subjects with significant cardio-vascular, pulmonary, renal, hepatic, gastro-intestinal, neurological, psychiatric, endocrine, cancer or blood disease,
14. Subjects having taken any unstable treatment with central effects within 90 days prior to experiment,
15. Subjects with an alcohol consumption more than 40 g of alcohol per day,
16. Subjects drinking more than 6 cups of coffee (or equivalent in xanthine-containing beverages) per day,
17. Subjects smoking more than 5 cigarettes per day,
18. Subjects with known drug addiction,
19. Subjects having donated more than 300 ml of blood within 90 days prior to the start of the study,
20. Subjects being in the exclusion period according to the French National File for Volunteers Participating in a Biomedical Research,
21. Subjects having earned a total annual amount of compensation from participating in clinical studies exceeding 4500 Euros (including compensation for this study),
22. Subjects with legal incapacity or limited legal capacity,
23. Subjects likely, according to investigator's opinion, not to cooperate with or to respect the constraints of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Number and description of participants with adverse events | 5 days
  adverse events will be recorded and reported throughout the study

SECONDARY OUTCOMES:
Neu-P11 concentration, exposure and clearance | 5 days
  To learn about the concentration, exposure and clearence of to Neu-P11 Pharmacokinetic(PK)parameters will be recorded and reported:
  * Blood samples for Neu-P11 and metabolites plasma concentration determination will be drawn on several time points at the beginning and at the end of each period
  * Urine samples for Neu-P11 and metabolites determination will be collected on several time points at the beginning and at the end of each period.
Objective and subjective assessment sleep quality | 5 days
  PSG parameters (sleep time, efficiency and architecture) as an objective assessment of sleep quality will be recorded
  Subjective means of evaluation of sleep qulity will include:
  * Sleep Diary (NSFSD).
  * sleepiness scale (KSS)
Subjective evaluation of mood and emotions | 5 days
  To study the effect of Neu-P11 on mood and emotions, subjective evaluation of mood and emotions will be recorded and reported using:
  * Profile of Mood States (POMS).
  * Emotional-visual analogue scale (e-VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Metzger, MD, Principal Investigator — Forenap Pharma
Locations (1):
- Centre hospitallier de Rouffach, Rouffach, France